CLINICAL TRIAL: NCT05128578
Title: Improving Pain Management and Opioid Safety for Patients With Cirrhosis: Pilot Program
Brief Title: Improving Pain Management and Opioid Safety for Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Shari Rogal, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21080148; 1K23DA048182-01A1 (NIH)
Record Dates: First submitted 2021-10-18; First posted 2021-11-22 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Cirrhosis, Liver
Keywords: liver diseases; cirrhosis, liver; implementation science; strategies; evaluation; behavioral intervention
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Intervention Model Description: LEAP is a modular 12-week pain self-management intervention with 6 individual sessions and 6 optional group sessions. Individual sessions serve the purpose of individualizing the program to the needs of the patients. Group sessions allow participants to practice skills, set goals with the group, seek social support, and learn together. The purpose of the LEAP program is to make pain better, help patients reach their personal goals (things that may be hard to do because of pain), and add to the care patients' medical team is providing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LEAP Intervention Arm (Experimental): Enrolled patients participated in weekly sessions led by a health coach to learn self-pain management tools and skills. There were 6 individual session and 6 optional group sessions. Participants also received an intervention manual with workbook activities they could complete.
  Interventions: Behavioral: Liver Education About Pain (LEAP); Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Liver Education About Pain (LEAP) — LEAP is a modular 12-week pain self-management intervention with 6 individual sessions and 6 optional group sessions. Individual sessions serve the purpose of individualizing the program to the needs of the patients. Group sessions allow participants to practice skills, set goals with the group, seek social support, and learn together. The purpose of the LEAP program is to make pain better, help patients reach their personal goals (things that may be hard to do because of pain), and add to the care patients' medical team is providing.
Behavioral: Usual Care — Patients can continue to use other pain management strategies ("usual care") in order to mimic real-life conditions.

SUMMARY:
This project aims to test a behavioral intervention in patients with liver cirrhosis and chronic pain and teach self pain-management skills.

DETAILED DESCRIPTION:
Prescription opioid medications are a leading cause of opioid-related death and are particularly risky in patients with cirrhosis of the liver, which affects 4 million people in the US. In this population, prescription opioids are associated with complications of liver disease, decreased access to life-saving transplantation, and increased hospitalization, post-transplant mortality, and all-cause mortality. Moreover, most patients with cirrhosis have underlying alcohol and/or substance use disorders (SUDs), which increase the risk of opioid-related complications and misuse. Despite these risks, our pilot work found that nearly half of all patients with cirrhosis are prescribed opioid medications each year and that these prescriptions are often inconsistent with opioid prescribing safety guidelines. One potential reason for this may be the lack of safe, evidence-based, alternative pain management strategies for this patient population. Indeed, existing opioid safety and pain management interventions designed for general populations do not address many of the specific issues facing patients with cirrhosis.

The research team plans to recruit patients at UPMC for participation in the Liver Education About Pain (LEAP) intervention program. LEAP is a modular 12-week pain self-management intervention with individual and group sessions. Individual sessions serve the purpose of individualizing the program to the needs of the patients. Group sessions allow participants to practice skills, set goals with the group, seek social support, and learn together. The purpose of the LEAP program is to make pain better, help patients reach their personal goals (things that may be hard to do because of pain), and add to the care patients' medical team is providing.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be over 18 years of age and fluent in English
* Must have a diagnosis of cirrhosis
* Must be receiving care at UPMC hepatology clinics
* Must have chronic pain lasting at least 3 months

Exclusion Criteria:

* Participants will be excluded if they are younger than 18 years of age or are unable to provide informed consent for any reason
* Participants will be excluded if they had a prior liver transplantation or have a limited life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2023-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari S Rogal, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited using fliers, mailings followed by calls, in-person clinic recruitment, and Pitt+Me, a service where potential participants can contact researchers for screening. The first participant was enrolled on March 14, 2022, and the last participant was enrolled in March 2023.
Groups:
- LEAP Intervention Arm: Enrolled patients will participate in 12 weekly sessions led by a health coach to learn self-pain management tools and skills. In addition to 6 individual sessions and 6 optional group sessions, participants will complete activities from the LEAP workbook (provided after enrollment), as tracking is a key component of most pain-self management interventions and is intended to address self-regulation. All patients can continue to use other pain management strategies ("usual care") in order to mimic real-life conditions.
  Liver Education About Pain (LEAP): LEAP is a modular 12-week pain self-management intervention with 6 individual sessions and 6 optional group sessions. Individual sessions serve the purpose of individualizing the program to the needs of the patients. Group sessions allow participants to practice skills, set goals with the group, seek social support, and learn together. The purpose of the LEAP program is to make pain better, help patients reach their personal goals (things that may be hard to do because of pain), and add to the care patients' medical team is providing.
  Usual Care: Patients can continue to use other pain management strategies ("usual care") in order to mimic real-life conditions.
Period: Overall Study
Arm/Group | LEAP Intervention Arm
Started | 30 (Enrolled in the study)
Baseline Survey | 24
Received Intervention | 21
Completed | 16 (Completed LEAP intervention)
Not Completed | 14
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: participants who started the intervention
Groups:
- LEAP Intervention Arm: Participants took part in Liver Education About Pain (LEAP), a modular, virtual 12-week pain self-management intervention. The 6 individual sessions and 6 optional group sessions were led by a health coach to help participants learn self-pain management tools and skills. Individual sessions served to tailor the program to the needs of the participants. Group sessions allowed participants to practice skills, set goals with the group, seek social support, and learn together. As part of the intervention, participants also received a manual ("LEAP manual") with useful information and activities to help with goal setting and tracking progress.
  Participants also continued to use any other pain management strategies ("usual care") in order to mimic real-life conditions.
Arm/Group | LEAP Intervention Arm
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  Overall: <=18 years | 0
  Overall: Between 18 and 65 years | 15
  Overall: >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years]
  Overall | 57.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Model for End-Stage Liver Disease (MELD) [Median (Inter-Quartile Range); unit: units on a scale] — This is a validated predictor of mortality among people with cirrhosis that is based on lab results and used across clinical care and research studies. THe scale is from 5-40, where a higher score represents worse outcome and more severe disease.
  units on a scale | 9 [7 to 11]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending ≥80% of Intervention Sessions
Description: participants who started intervention and completed ≥80% of intervention sessions divided by the number who started intervention (completed a session)
Time Frame: post intervention (6 months)
Population: number of participant who completed at least 80% of sessions/Participants who started intervention
Measure: Count of Participants; unit: Participants
Arm/Group | LEAP Intervention Arm
Number analyzed (Participants) | 21
Participants
  Completed 80% of sessions | 16
  Did not complete | 5

2. Primary Outcome: Overall Satisfaction
Description: Treatment expectations questionnaire (TEQ) was used to assess patient satisfaction. This is a 5-item, validated questionnaire includes Likert scale items on a 5-point scale from negative to positive views of different aspects of the intervention (-2 is highly negative views to +2 is highly positive views of the intervention). There is an option for I don't know. Primary outcome was measured using a mean of the mean scores on this Likert scale, where 1 is a somewhat positive view of the intervention and +2 is a highly positive view of the intervention.
Time Frame: end of intervention
Population: 12 patients completed this measure at the end of intervention. Note-one patient responded that they did not know about the intervention and was removed from further analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LEAP Intervention Arm
Number analyzed (Participants) | 12
units on a scale | 1.56 (.27)

ADVERSE EVENTS:
Time Frame: 6 months after the start of the intervention
Arm/Group | LEAP Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/78/NCT05128578/Prot_SAP_000.pdf